CLINICAL TRIAL: NCT03146351
Title: The Effects of Family Centered Physiotherapy Program on Preterm Infants
Brief Title: The Effects of Family Centered Intervention Program on Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Murat Fatih KOCYIGIT, Research Assistant, Gazi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MURATKOCYİGİT
Record Dates: First submitted 2017-04-19; First posted 2017-05-09 (Actual); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Infant, Premature
Keywords: preterm; infant; physiotherapy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: non-randomised clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early and moderate preterm group (Experimental): Infants born before 34 weeks included in this group
  Interventions: Other: Family based early intervention program (NDT-Bobath based)
- Late preterm group (Experimental): Infants born between 34 and 37 weeks included in this group
  Interventions: Other: Family based early intervention program (NDT-Bobath based)

INTERVENTIONS:
Other: Family based early intervention program (NDT-Bobath based) — Family based early intervention program is NDT - Bobath based home program. Physiotherapist teaches principles of the treatment to infants' family. Family applies the program at home.

SUMMARY:
Infant born preterm have an increased risk of adverse long-term developmental outcomes.The risk associated with preterm birth increase as gestational age decreases, and vulnerability remains in moderate and early preterm (<34 weeks) and late preterm (>34 weeks). There are many studies in the literature showed that the prevalence of developmental delay increases with premature birth. However, there is no study in the literature investigates effect of early intervention program motor performance in subgroups of preterm infants. Hence the aim of this study is to evaluate the differences in effects of early intervention program on motor development in early and moderate (<34 weeks) and late preterm infants.

DETAILED DESCRIPTION:
Fifty-two preterm infants corrected age less than 6 months included in this study. They were separated by their birth weeks. Babies with gestational ages between 34-36 weeks and 6 days (including the given days) are categorized as late preterm, while those born before 34 weeks are grouped as moderate and early preterm. Each group contains 26 infants.

First, sociodemographic information and histories of babies are obtaining. Ages and contact information of the parents are recording. Prenatal and natal risk factors of the mothers are querying. Gestational ages and height, weight, and head circumferences of babies at birth are recording. Number of pregnancies, live births and abortions, type of delivery, multiple pregnancies for mothers as well as consanguinity between parents are asking.The Alberta Infant Motor Scale is using to evaluate spontaneous motor movements of the baby. After the detailed examination, intervention program set up for infants. Both groups receive 3 months family based intervention program.

After the intervention program, both groups re-examined.

ELIGIBILITY:
Inclusion Criteria:

* Born before 37 gestational weeks,
* Accepting to join the study
* Corrected age 6 months or less

Exclusion Criteria:

* Having high risk factors (e.g. grade 3 or more intraventricular hemorrhage, PVL, serious seizure)
* Born after 37 weeks
* Corrected age greater than 6 months

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Motor performance using the Alberta Infant Motor Scale | This study is planned to be completed within 6 months
  Alberta Infant Motor Scale is used to examine motor performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi Universitesi, Saglik Bilimleri Fakultesi, Fizyoterapi ve Rehabilitasyon Bolumu, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We have no decided yet

REFERENCES:
- [Background] Kyno NM, Ravn IH, Lindemann R, Fagerland MW, Smeby NA, Torgersen AM. Effect of an early intervention programme on development of moderate and late preterm infants at 36 months: a randomized controlled study. Infant Behav Dev. 2012 Dec;35(4):916-26. doi: 10.1016/j.infbeh.2012.09.004. Epub 2012 Oct 11. PMID 23063851